CLINICAL TRIAL: NCT06645990
Title: Early Left Ventricular unLoading by Impella (ECMELLA) or Intra-aortic Balloon Pump for Cardiogenic Shock in Patients on VA-ECMO
Brief Title: Early Left Ventricular unLoading by Impella vs Intra-aortic Balloon Pump
Acronym: ELLIPSE1
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-06-079
Record Dates: First submitted 2024-10-01; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Cardiogenic Shock
Keywords: ECMO; ECLS; Impella; IABP; pVAD; mortality
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ECMELLA group: VA-ECMO + Impella implemented before or within 24 h of ECMO initiation
  Interventions: Device: Impella
- ECMO+IABP group: VA-ECMO + IABP implemented before or within 24h of ECMO initiation
  Interventions: Device: IABP

INTERVENTIONS:
Device: Impella — LV unloading with Impella (ECMELLA) before or within 24 h of ECMO initiation
  Groups: ECMELLA group
Device: IABP — LV unloading with IABP before or within 24 h of ECMO initiation
  Groups: ECMO+IABP group

SUMMARY:
Over the past decade, VA-ECMO has become the main mechanical support for cardiogenic shock (CS) unresponsive to medical therapy. However, recent studies failed to show any significant survival benefit at 30 days compared to medical treatment for myocardial infarction-related CS. This could be due to the complications of VA-ECMO, such as LV overload and increased LV distension, which can hinder heart recovery.

To address this, early LV unloading using devices like IABP or Impella (ECMELLA) may help by reducing LV wall stress and oxygen consumption. However, these techniques carry risks, and their benefit is still unclear. A randomized trial is needed to compare these approaches, but observational studies are also contributing to understanding the best strategies

DETAILED DESCRIPTION:
Over the last decade, veno-arterial extracorporeal membrane oxygenation (VA-ECMO) has become the mechanical circulatory support of choice for cardiogenic shock (CS) refractory to medical treatment. VA-ECMO allows to supplement cardiac function until myocardium recovers, or in bridge to long-term left ventricular assist device (LVAD) or to heart transplant. However, recent randomized controlled trials (RCT) and meta-analysis have failed to demonstrate any benefit of VA-ECMO in terms of 30-day survival compared with optimal medical treatment in CS related to myocardial infarction.

Reasons for these disappointing results are multifactorial. The associated risk of temporary mechanical circulatory support (t-MCS)-related complications might counterbalance any hemodynamic benefit. In addition to hemorrhagic and ischemic complications, the significant myocardial impact due to VA-ECMO drawbacks should not be overlooked. Indeed, while VA-ECMO restores systemic perfusion, it can also lead to an increase in left ventricle (LV) loading conditions. Although LV distension is not consistently observed, recent publications strongly suggest that the origin of LV overload seems to be multifactorial and contributes partially to cardiac remodeling through the modulation of cardioprotective cellular pathways, resulting in reduced cardiomyocyte apoptosis. Furthermore, peripheral VA-ECMO affects myocardial contractility and increases myocardial work (potential energy, stroke work, and pressure-volume area), particularly at native low blood flow.

Thus, cardiac recovery may be compromised and weaning from VA-ECMO delayed. This vicious cycle affects the patients overall prognosis, as delayed and possibly failure of VA-ECMO weaning and may convert the initial medical strategy of recovery towards heart transplantation or LVAD. To optimize the chance of VA-ECMO weaning, early LV unloading may be a good therapeutic option. It aims at increasing coronary flow directly and, indirectly, by improving sub-endocardial myocardial perfusion through decreasing LV wall stress and myocardial oxygen consumption. Currently, 2 techniques are mainly used, the intra-aortic balloon pump (IABP) and the microaxial flow pump as Impella device familly (ECMELLA). These invasive techniques carry risks of bleeding and thromboembolic complications, and the benefit/risk ratio of their use for myocardial recovery is not clearly established.

A few retrospective studies suggest that early left ventricular unloading during VA-ECMO could improve prognosis. In the absence of RCT, the choice of the technique (Impella or IABP) is mainly driven by center practice. A multicenter randomized clinical trial would be the best choice to address this question. However, due to the acute poor prognosis of these patients (50% of early deaths), reliable preliminary data about the expected effect size are necessary to design the most efficient clinical trial. Recent epidemiologic developments of observational studies, the emulated trials, allow a better control of immortal time bias and indication bias.

This innovative multicenter study will compare the effectiveness and safety of LV unloading by Impella (ECMELLA) versus IABP in terms of survival with myocardial recovery in patients with refractory CS

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (more than or =18 years) admitted for cardiogenic shock supported by ECMO+ IABP or ECMELLA between January 1, 2010, and December 31, 2023

Exclusion Criteria:

* Ongoing extra-corporeal CardioPulmonary Resuscitation (eCPR) at time of ECMO implantation
* Cardiogenic shock with previous prolonged continuous cardiopulmonary resuscitation (CPR) more than 30 minutes
* Acute irreversible neurological injury
* Previous known severe chronic cardiomyopathy (LVEF less than 25%) or awaiting heart transplantation or LVAD implantation
* Contraindication to the implantation of an Impella or IABP
* Mechanical complications of myocardial infarction
* Moribund patient (SAPS more than 90)
* Previous known severe chronic renal or hepatic failure
* Age less than18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Adult patients (more than or =18 years) admitted for Cardiogenic Shock supported by ECMO+ IABP or ECMELLA between January 1, 2010, and December 31, 2023
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Myocardial recovery | from start of hospitalization until hospital discharge assessed up to 3 month
  Hospital Survival without chronic mechanical circulatory support (LVAD) and heart transplantation.

SECONDARY OUTCOMES:
Early mortality | from start of hospitalization until hospital discharge assessed up to 3 month
  In-hospital all-cause mortality
Adverse events related to LV unloading technics | from start of hospitalization until hospital discharge assessed up to 3 month
  Arterial thromboembolic events; Hemorrhagic events (RBC transfusion); Hemolysis; Bacteremia; Infection of the device insertion site or the device itself
Duration of mechanical ventilation | from start of hospitalization until hospital discharge assessed up to 3 month
  Total duration of invasive mechanical ventilation
Duration of temporary MCS support | from start of hospitalization until hospital discharge assessed up to 3 month
  Total duration of t-MCS
Lengh of stay | from start of hospitalization until hospital discharge assessed up to 3 month
  Total and in intensive care unit lenght of stay
Cardiac long-term project | from start of hospitalization until hospital discharge assessed up to 3 month
  Rate and % of patients with myocardial recovery, ventricular assist device or/and heart transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Aurore UGHETTO, MD, Principal Investigator — Montpellier University Hospital, France
Locations (1):
- CHU Arnaud de Villeneuve, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Authors/Task Force Members:; McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: Developed by the Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC). With the special contribution of the Heart Failure Association (HFA) of the ESC. Eur J Heart Fail. 2022 Jan;24(1):4-131. doi: 10.1002/ejhf.2333. PMID 35083827
- [Background] Pocock SJ, Ariti CA, Collier TJ, Wang D. The win ratio: a new approach to the analysis of composite endpoints in clinical trials based on clinical priorities. Eur Heart J. 2012 Jan;33(2):176-82. doi: 10.1093/eurheartj/ehr352. Epub 2011 Sep 6. PMID 21900289
- [Background] Hernan MA, Sauer BC, Hernandez-Diaz S, Platt R, Shrier I. Specifying a target trial prevents immortal time bias and other self-inflicted injuries in observational analyses. J Clin Epidemiol. 2016 Nov;79:70-75. doi: 10.1016/j.jclinepi.2016.04.014. Epub 2016 May 27. PMID 27237061
- [Background] Hernan MA, Robins JM. Using Big Data to Emulate a Target Trial When a Randomized Trial Is Not Available. Am J Epidemiol. 2016 Apr 15;183(8):758-64. doi: 10.1093/aje/kwv254. Epub 2016 Mar 18. PMID 26994063
- [Background] Ezad SM, Ryan M, Donker DW, Pappalardo F, Barrett N, Camporota L, Price S, Kapur NK, Perera D. Unloading the Left Ventricle in Venoarterial ECMO: In Whom, When, and How? Circulation. 2023 Apr 18;147(16):1237-1250. doi: 10.1161/CIRCULATIONAHA.122.062371. Epub 2023 Apr 17. PMID 37068133
- [Background] Bernhardt AM, Copeland H, Deswal A, Gluck J, Givertz MM; Chairs:; Co-Chairs:; Contributing Writers:; Chair:; Co-Chair:; Contributing Writers:; Chair:; Co-Chairs:; Contributing Writers:; Chair:; Co-Chair:; Contributing Writers:. The International Society for Heart and Lung Transplantation/Heart Failure Society of America Guideline on Acute Mechanical Circulatory Support. J Heart Lung Transplant. 2023 Apr;42(4):e1-e64. doi: 10.1016/j.healun.2022.10.028. Epub 2023 Feb 6. No abstract available. PMID 36805198
- [Result] Ostadal P, Rokyta R, Karasek J, Kruger A, Vondrakova D, Janotka M, Naar J, Smalcova J, Hubatova M, Hromadka M, Volovar S, Seyfrydova M, Jarkovsky J, Svoboda M, Linhart A, Belohlavek J; ECMO-CS Investigators. Extracorporeal Membrane Oxygenation in the Therapy of Cardiogenic Shock: Results of the ECMO-CS Randomized Clinical Trial. Circulation. 2023 Feb 7;147(6):454-464. doi: 10.1161/CIRCULATIONAHA.122.062949. Epub 2022 Nov 6. PMID 36335478
- [Result] Banning AS, Sabate M, Orban M, Gracey J, Lopez-Sobrino T, Massberg S, Kastrati A, Bogaerts K, Adriaenssens T, Berry C, Erglis A, Haine S, Myrmel T, Patel S, Buera I, Sionis A, Vilalta V, Yusuff H, Vrints C, Adlam D, Flather M, Gershlick AH. Venoarterial extracorporeal membrane oxygenation or standard care in patients with cardiogenic shock complicating acute myocardial infarction: the multicentre, randomised EURO SHOCK trial. EuroIntervention. 2023 Aug 21;19(6):482-492. doi: 10.4244/EIJ-D-23-00204. PMID 37334659
- [Result] Thiele H, Zeymer U, Akin I, Behnes M, Rassaf T, Mahabadi AA, Lehmann R, Eitel I, Graf T, Seidler T, Schuster A, Skurk C, Duerschmied D, Clemmensen P, Hennersdorf M, Fichtlscherer S, Voigt I, Seyfarth M, John S, Ewen S, Linke A, Tigges E, Nordbeck P, Bruch L, Jung C, Franz J, Lauten P, Goslar T, Feistritzer HJ, Poss J, Kirchhof E, Ouarrak T, Schneider S, Desch S, Freund A; ECLS-SHOCK Investigators. Extracorporeal Life Support in Infarct-Related Cardiogenic Shock. N Engl J Med. 2023 Oct 5;389(14):1286-1297. doi: 10.1056/NEJMoa2307227. Epub 2023 Aug 26. PMID 37634145
- [Result] Schmidt M, Burrell A, Roberts L, Bailey M, Sheldrake J, Rycus PT, Hodgson C, Scheinkestel C, Cooper DJ, Thiagarajan RR, Brodie D, Pellegrino V, Pilcher D. Predicting survival after ECMO for refractory cardiogenic shock: the survival after veno-arterial-ECMO (SAVE)-score. Eur Heart J. 2015 Sep 1;36(33):2246-56. doi: 10.1093/eurheartj/ehv194. Epub 2015 Jun 1. PMID 26033984
- [Result] Muller G, Flecher E, Lebreton G, Luyt CE, Trouillet JL, Brechot N, Schmidt M, Mastroianni C, Chastre J, Leprince P, Anselmi A, Combes A. The ENCOURAGE mortality risk score and analysis of long-term outcomes after VA-ECMO for acute myocardial infarction with cardiogenic shock. Intensive Care Med. 2016 Mar;42(3):370-378. doi: 10.1007/s00134-016-4223-9. Epub 2016 Jan 29. PMID 26825953
- [Result] Dickerman BA, Garcia-Albeniz X, Logan RW, Denaxas S, Hernan MA. Avoidable flaws in observational analyses: an application to statins and cancer. Nat Med. 2019 Oct;25(10):1601-1606. doi: 10.1038/s41591-019-0597-x. Epub 2019 Oct 7. PMID 31591592
- [Result] Meuwese CL, Koudstaal S, Braithwaite S, Hermens JAJ, Donker DW. Left Ventricular Unloading During Extracorporeal Membrane Oxygenation: Insights From Meta-Analyzed Observational Data Corrected for Confounders. J Am Coll Cardiol. 2019 Jun 18;73(23):3034-3035. doi: 10.1016/j.jacc.2019.03.505. No abstract available. PMID 31196464
- [Result] Beurton A, Michot M, Herion FX, Rienzo M, Oddos C, Couffinhal T, Imbault J, Ouattara A. Systemic Hemodynamics, Cardiac Mechanics, and Signaling Pathways Induced by Extracorporeal Membrane Oxygenation in a Cardiogenic Shock Model. ASAIO J. 2024 Mar 1;70(3):177-184. doi: 10.1097/MAT.0000000000002139. Epub 2024 Jan 23. PMID 38261663
- [Result] Ughetto A, Eliet J, Nagot N, David H, Bazalgette F, Marin G, Kollen S, Mourad M, Zeroual N, Muller L, Gaudard P, Colson P. Early temporary mechanical circulatory support for cardiogenic shock: Real-life data from a regional cardiac assistance network. J Heart Lung Transplant. 2024 Jun;43(6):911-919. doi: 10.1016/j.healun.2024.02.009. Epub 2024 Feb 15. PMID 38367739